CLINICAL TRIAL: NCT02325713
Title: A Phase I, Open-label, Randomized, Four-period, Crossover, Single Center Trial to Assess the Relative Bioavailability of a Single Oral Dose of the New 150 mg Oral Dispersible Tablet (ODT) Formulation of Praziquantel (PZQ), MSC1028703A, at Different Dose Levels vs the Current Commercial 500 mg Tablet Formulation of PZQ in Healthy Male Volunteers
Brief Title: Relative Bioavailability Trial of Oral Dispersible Praziquantel Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200585-001
Record Dates: First submitted 2014-12-11; First posted 2014-12-25 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Healthy
Keywords: ODT-PZQ; Bio-availability; Praziquantel; Cysticide; Pharmacokinetics
MeSH Terms: interventions — Praziquantel

ARMS (16):
- Sequence A-B-C1-D1 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence A-B-C1-D2 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence A-B-C2-D1 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence A-B-C2-D2 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence A-B-D1-C1 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence A-B-D2-C1 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence A-B-D1-C2 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence A-B-D2-C2 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence B-A-C1-D1 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence B-A-C1-D2 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence B-A-C2-D1 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence B-A-C2-D2 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence B-A-D1-C1 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence B-A-D2-C1 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence B-A-D1-C2 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ
- Sequence B-A-D2-C2 (Experimental)
  Interventions: Drug: Oral dispersible tablet of praziquantel (ODT-PZQ); Drug: Cysticide; Drug: ODT-PZQ

INTERVENTIONS:
Drug: Oral dispersible tablet of praziquantel (ODT-PZQ) — Treatment A (test): ODT-PZQ (MSC1028703A) at a single dose of 40 milligram per kilogram (mg/kg) orally dispersed in water after meal.
  Other Names: MSC1028703A
Drug: Cysticide — Treatment B (reference): Cysticide tablet at a single dose of 40 mg/kg will be given with water orally after a meal.
  Other Names: PZQ
Drug: ODT-PZQ — Treatment C1 (test): ODT-PZQ (MSC1028703A) at a single dose of 20 mg/kg orally dispersed in water after a meal.
  Other Names: MSC1028703A
  Arms: Sequence A-B-C1-D1; Sequence A-B-C1-D2; Sequence A-B-D1-C1; Sequence A-B-D2-C1; Sequence B-A-C1-D1; Sequence B-A-C1-D2; Sequence B-A-D1-C1; Sequence B-A-D2-C1
Drug: ODT-PZQ — Treatment C2 (test): ODT-PZQ (MSC1028703A) at a single dose of 60 mg/kg orally dispersed in water after a meal.
  Other Names: MSC1028703A
  Arms: Sequence A-B-C2-D1; Sequence A-B-C2-D2; Sequence A-B-D1-C2; Sequence A-B-D2-C2; Sequence B-A-C2-D1; Sequence B-A-C2-D2; Sequence B-A-D1-C2; Sequence B-A-D2-C2
Drug: ODT-PZQ — Treatment D1 (test): ODT-PZQ (MSC1028703A) at a single dose of 40 mg/kg orally dispersed in water without a meal.
  Other Names: MSC1028703A
  Arms: Sequence A-B-C1-D1; Sequence A-B-C2-D1; Sequence A-B-D1-C1; Sequence A-B-D1-C2; Sequence B-A-C1-D1; Sequence B-A-C2-D1; Sequence B-A-D1-C1; Sequence B-A-D1-C2
Drug: Cysticide — Treatment D2 (reference): Cysticide crushed tablets at a single dose of 40 mg/kg will be given with water orally after a meal.
  Other Names: PZQ
  Arms: Sequence A-B-C1-D2; Sequence A-B-C2-D2; Sequence A-B-D2-C1; Sequence A-B-D2-C2; Sequence B-A-C1-D2; Sequence B-A-C2-D2; Sequence B-A-D2-C1; Sequence B-A-D2-C2

SUMMARY:
This is a phase I, open-label, randomized, 4 period, crossover, single-center trial. The purpose of this trial is to assess the relative bio-availability of racemate Oral Dispersible Tablet praziquantel (ODT-PQZ) (MSC1028703A) 150 milligram (mg) versus the current marketed praziquantel (PZQ) (Cysticide® 500 mg) formulation in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males 18-55 years of age (inclusive at screening)
* Male subjects with partners of childbearing potential must have had a vasectomy or use acceptable methods of birth control (that is, condoms) and not donate sperm during, and until 90 days after the last dose of the trial medication
* Provide written informed consent prior to any trial related procedure
* Body weight of greater than or equal to (>=)55.0 kg to less than (<) 95.0 kg and a body mass index (BMI) between 18.5 and 29.9 kilogram per square meter (kg/m^2)
* Able to communicate well with the Investigator, understand the protocol requirements and restrictions, and willing to comply with the requirements of the entire trial
* Non-smoker (= 0 cigarettes, pipes, cigars or other) from at least 3 months prior to start of trial
* Electrocardiogram (ECG) recording (12-lead) without signs of clinically relevant pathology, in particular QTcB < 450 milliseconds (ms)
* Vital signs (systolic blood pressure, diastolic blood pressure and pulse) in supine position are within the normal range or show no clinically relevant deviation as judged by the Investigator

Exclusion Criteria:

* Any surgical or medical condition, including findings in the medical history or in the pre-study assessments, or any other significant disease, that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the subject in the trial or that could interfere with the trial objectives, conduct or evaluation
* History of gastrointestinal (GI) tract surgery, other GI tract diseases or acute GI tract infections within the last 2 weeks that could influence the GI absorption and/or motility according to the Investigator's opinion
* Any clinically relevant abnormality in the safety laboratory parameters as judged by the Investigator
* Positive results from serology examination for Hepatitis B surface antigen (HBsAg), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV)
* Have an ascertained or presumptive contraindication or hypersensitivity to the active drug substance and/or formulations' ingredients
* Have any clinically significant history of allergic conditions which the Investigator considers may affect the outcome of the trial
* History or presence of drug abuse or alcohol abuse (as defined by the assessment of the investigator) at screening and on each admission
* Blood donation or loss of more than 400 mL of blood within 3 months before the first administration of the investigational product
* Administration of any investigational product or use of any investigational device within 60 days prior to first dosing that may affect the pharmacokinetics of the investigational product
* Subjects who have used drugs that may affect the pharmacokinetics (PK) of PZQ from 15 days before the first administration of the investigational product until the last PK sample
* Consumption of substances known to be potent inhibitors or inducers of cytochrome P450s (CYPs) within 2 weeks before the first administration of the investigational product
* Unlikely to comply with the protocol requirements, instructions and trial-related restrictions
* Non-acceptance of the study breakfast
* Excessive consumption of beverages containing xanthine (greater than [>] 5 cups of coffee a day or equivalent) and the inability to refrain from the use of caffeine-containing beverages from 48 hours before the first administration of the investigational product until discharge from the clinic
* Subject is the Investigator or any Sub-Investigator, research assistant, pharmacist, trial coordinator, other staff or relative thereof directly involved in the conduct of the trial
* Vulnerable subjects
* Legal incapacity or limited legal capacity

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last subject (informed consent): 21 January 2015/21 January 2015. Study completion date: 09 March 2015. The study was conducted at one center in South Africa.
Pre-assignment Details: Overall, 65 subjects were screened, for inclusion in this trial. Of which, 32 subjects were enrolled and randomized to a treatment sequence.
Groups:
- Sequence A-B-C1-D1: Subjects randomized to treatment sequence A-B-C1-D1 received a single oral dose of 40 milligram per kilogram (40 mg/kg) of test oral dispersible tablet of praziquantel (ODT-PZQ) dispersed in water after a meal (Treatment A) in first intervention period and then reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in second intervention period and then a single oral dose 20 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C1) in third intervention period and then a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water without a meal (Treatment D1) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence A-B-C1-D2: Subjects randomized to treatment sequence A-B-C1-D2 received a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in first intervention period and then reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in second intervention period and then a single oral dose 20 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C1) in third intervention period and then reference PZQ formulation (Cysticide crushed tablets) at a single dose of 40 mg/kg given with water orally after a meal (Treatment D2) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence A-B-C2-D1: Subjects randomized to treatment sequence A-B-C2-D1 received a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in first intervention period and then reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in second intervention period and then a single oral dose 60 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C2) in third intervention period and then a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water without a meal (Treatment D1) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence A-B-C2-D2: Subjects randomized to treatment sequence A-B-C2-D2 received a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in first intervention period and then reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in second intervention period and then a single oral dose 60 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C2) in third intervention period and then reference PZQ formulation (Cysticide crushed tablets) at a single dose of 40 mg/kg given with water orally after a meal (Treatment D2) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence A-B-D1-C1: Subjects randomized to treatment sequence A-B-D1-C1 received a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in first intervention period and then reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in second intervention period and then a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water without a meal (Treatment D1) in third intervention period and then a single oral dose 20 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C1) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence A-B-D2-C1: Subjects randomized to treatment sequence A-B-D2-C1 received a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in first intervention period and then reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in second intervention period and then reference PZQ formulation (Cysticide crushed tablets) at a single dose of 40 mg/kg given with water orally after a meal (Treatment D2) in third intervention period and then a single oral dose 20 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C1) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence A-B-D1-C2: Subjects randomized to treatment sequence A-B-D1-C2 received a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in first intervention period and then reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in second intervention period and then a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water without a meal (Treatment D1) in third intervention period and then a single oral dose 60 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C2) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence A-B-D2-C2: Subjects randomized to treatment sequence A-B-D2-C2 received a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in first intervention period and then reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in second intervention period and then reference PZQ formulation (Cysticide crushed tablets) at a single dose of 40 mg/kg given with water orally after a meal (Treatment D2) in third intervention period and then a single oral dose 60 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C2) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence B-A-C1-D1: Subjects randomized to treatment sequence B-A-C1-D1 received reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in first intervention period and then a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in second intervention period and then a single oral dose 20 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C1) in third intervention period and then a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water without a meal (Treatment D1) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence B-A-C1-D2: Subjects randomized to treatment sequence B-A-C1-D2 received reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in first intervention period and then a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in second intervention period and then a single oral dose 20 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C1) in third intervention period and then reference PZQ formulation (Cysticide crushed tablets) at a single dose of 40 mg/kg given with water orally after a meal (Treatment D2) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence B-A-C2-D1: Subjects randomized to treatment sequence B-A-C2-D1 received reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in first intervention period and then a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in second intervention period and then a single oral dose 60 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C2) in third intervention period and then a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water without a meal (Treatment D1) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence B-A-C2-D2: Subjects randomized to treatment sequence B-A-C2-D2 received reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in first intervention period and then a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in second intervention period and then a single oral dose 60 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C2) in third intervention period and then reference PZQ formulation (Cysticide crushed tablets) at a single dose of 40 mg/kg given with water orally after a meal (Treatment D2) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence B-A-D1-C1: Subjects randomized to treatment sequence B-A-D1-C1 received reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in first intervention period and then a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in second intervention period and then a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water without a meal (Treatment D1) in third intervention period and then a single oral dose 20 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C1) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence B-A-D2-C1: Subjects randomized to treatment sequence B-A-D2-C1 received reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in first intervention period and then a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in second intervention period and then reference PZQ formulation (Cysticide crushed tablets) at a single dose of 40 mg/kg given with water orally after a meal (Treatment D2) in third intervention period and then a single oral dose 20 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C1) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence B-A-D1-C2: Subjects randomized to treatment sequence B-A-D1-C2 received reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in first intervention period and then a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in second intervention period and then a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water without a meal (Treatment D1) in third intervention period and then a single oral dose 60 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C2) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
- Sequence B-A-D2-C2: Subjects randomized to treatment sequence B-A-D2-C2 received reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal (Treatment B) in first intervention period and then a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment A) in second intervention period and then reference PZQ formulation (Cysticide crushed tablets) at a single dose of 40 mg/kg given with water orally after a meal (Treatment D2) in third intervention period and then a single oral dose 60 mg/kg of test ODT-PZQ dispersed in water after a meal (Treatment C2) in fourth intervention period. A washout period of 7 days was maintained between each intervention period.
Period: Intervention Period 1 (2 Days)
Arm/Group | Sequence A-B-C1-D1 | Sequence A-B-C1-D2 | Sequence A-B-C2-D1 | Sequence A-B-C2-D2 | Sequence A-B-D1-C1 | Sequence A-B-D2-C1 | Sequence A-B-D1-C2 | Sequence A-B-D2-C2 | Sequence B-A-C1-D1 | Sequence B-A-C1-D2 | Sequence B-A-C2-D1 | Sequence B-A-C2-D2 | Sequence B-A-D1-C1 | Sequence B-A-D2-C1 | Sequence B-A-D1-C2 | Sequence B-A-D2-C2
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Non-Compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 2 (2 Days)
Arm/Group | Sequence A-B-C1-D1 | Sequence A-B-C1-D2 | Sequence A-B-C2-D1 | Sequence A-B-C2-D2 | Sequence A-B-D1-C1 | Sequence A-B-D2-C1 | Sequence A-B-D1-C2 | Sequence A-B-D2-C2 | Sequence B-A-C1-D1 | Sequence B-A-C1-D2 | Sequence B-A-C2-D1 | Sequence B-A-C2-D2 | Sequence B-A-D1-C1 | Sequence B-A-D2-C1 | Sequence B-A-D1-C2 | Sequence B-A-D2-C2
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2
Completed | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Non-Compliance | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 3 (2 Days)
Arm/Group | Sequence A-B-C1-D1 | Sequence A-B-C1-D2 | Sequence A-B-C2-D1 | Sequence A-B-C2-D2 | Sequence A-B-D1-C1 | Sequence A-B-D2-C1 | Sequence A-B-D1-C2 | Sequence A-B-D2-C2 | Sequence B-A-C1-D1 | Sequence B-A-C1-D2 | Sequence B-A-C2-D1 | Sequence B-A-C2-D2 | Sequence B-A-D1-C1 | Sequence B-A-D2-C1 | Sequence B-A-D1-C2 | Sequence B-A-D2-C2
Started | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2
Completed | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 4 (2 Days)
Arm/Group | Sequence A-B-C1-D1 | Sequence A-B-C1-D2 | Sequence A-B-C2-D1 | Sequence A-B-C2-D2 | Sequence A-B-D1-C1 | Sequence A-B-D2-C1 | Sequence A-B-D1-C2 | Sequence A-B-D2-C2 | Sequence B-A-C1-D1 | Sequence B-A-C1-D2 | Sequence B-A-C2-D1 | Sequence B-A-C2-D2 | Sequence B-A-D1-C1 | Sequence B-A-D2-C1 | Sequence B-A-D1-C2 | Sequence B-A-D2-C2
Started | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 2
Completed | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized subjects who received at least 1 dose of the trial medication and who had follow-up safety assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A-B-C1-D1 | Sequence A-B-C1-D2 | Sequence A-B-C2-D1 | Sequence A-B-C2-D2 | Sequence A-B-D1-C1 | Sequence A-B-D2-C1 | Sequence A-B-D1-C2 | Sequence A-B-D2-C2 | Sequence B-A-C1-D1 | Sequence B-A-C1-D2 | Sequence B-A-C2-D1 | Sequence B-A-C2-D2 | Sequence B-A-D1-C1 | Sequence B-A-D2-C1 | Sequence B-A-D1-C2 | Sequence B-A-D2-C2 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 32

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUC0-inf) Adjusted for the Actual Administered Dose (AUC0-inf, Adj) of L-Praziquantel (L-PZQ)
Description: AUC0-inf is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time. AUC0-inf, adj was defined as the AUC0-inf adjusted for the actual administered dose of L-PZQ.
Time Frame: Pre-dose,0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: The pharmacokinetic (PK) population included all subjects who completed the study and for whom primary PK parameters could be calculated for the first two treatment periods. Here, 'N' (number of participants analyzed) signifies those subjects who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter (h*ng/mL)
Groups:
- Treatment A: 40 mg/kg Test ODT-PZQ After Meal: Subjects who received a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal in either of the four intervention periods.
- Treatment B: 40 mg/kg Cysticide Tablet After Meal: Subjects who received reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal either of the four intervention periods.
- Treatment C1: 20 mg/kg Test ODT-PZQ After Meal: Subjects who received a single oral dose of 20 mg/kg of test ODT-PZQ dispersed in water after a meal in either of the four intervention periods.
- Treatment C2: 60 mg/kg Test ODT-PZQ After Meal: Subjects who received a single oral dose 60 mg/kg of test ODT-PZQ dispersed in water after a meal in either of the four intervention periods.
- Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal: Subjects who received a single oral dose 40 mg/kg of test ODT-PZQ dispersed in water without a meal in either of the four intervention periods.
- Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal: Subjects who received reference PZQ formulation (Cysticide crushed tablets) at a single dose of 40 mg/kg given with water orally after a meal in either of the four intervention periods.
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 14 | 15 | 14 | 14
Hour*nanograms per milliliter (h*ng/mL) | 1969.6 (47.2) | 2047.9 (60.2) | 345.4 (69.5) | 4871.3 (42.2) | 924.9 (67.7) | 1537.7 (70.6)
Statistical Analysis 1: Comparison: Treatment A: 40 mg/kg Test ODT-PZQ After Meal vs Treatment B: 40 mg/kg Cysticide Tablet After Meal; Test type: Superiority or Other; Geometric Least square (LS) mean ratio = 96.2, 90% CI 2-sided [83.7 to 110.6]
Statistical Analysis 2: Comparison: Treatment A: 40 mg/kg Test ODT-PZQ After Meal vs Treatment C1: 20 mg/kg Test ODT-PZQ After Meal; Test type: Superiority or Other; Geometric LS mean ration = 18.4, 90% CI 2-sided [15.3 to 22.0]
Statistical Analysis 3: Comparison: Treatment A: 40 mg/kg Test ODT-PZQ After Meal vs Treatment C2: 60 mg/kg Test ODT-PZQ After Meal; Test type: Superiority or Other; Geometric LS mean ration = 222.7, 90% CI 2-sided [186.8 to 265.6]
Statistical Analysis 4: Comparison: Treatment A: 40 mg/kg Test ODT-PZQ After Meal vs Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal; Test type: Superiority or Other; Geometric LS mean ration = 238.1, 90% CI 2-sided [198.7 to 285.3]
Statistical Analysis 5: Comparison: Treatment B: 40 mg/kg Cysticide Tablet After Meal vs Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal; Test type: Superiority or Other; Geometric LS mean ration = 82.1, 90% CI 2-sided [68.5 to 98.3]

2. Secondary Outcome: Maximum Observed Concentration in Plasma (Cmax) Adjusted for the Actual Administered Dose (Cmax, Adj) of L-PZQ, D-PZQ and Racemate PZQ
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: The PK population included all subjects who completed the study and for whom primary PK parameters could be calculated for the first two treatment periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 14 | 15
ng/mL
  L-PZQ | 881.3 (57.2) | 762.6 (59.5) | 154.6 (80.4) | 1548 (32.6) | 189.3 (104.0) | 446.3 (87.6)
  D-PZQ | 2330 (30.7) | 2179 (33.0) | 786.3 (41.5) | 3234 (20.0) | 838.5 (65.7) | 1556 (35.8)
  Racemate PZQ | 3250 (34.6) | 2974 (37.2) | 949.9 (45.1) | 4780 (23.3) | 1042 (70.7) | 2040 (40.9)

3. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of L-PZQ, D-PZQ, and Racemate PZQ
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 14 | 15
hours
  L-PZQ | 3.000 [1.00 to 4.50] | 1.500 [1.00 to 4.50] | 4.000 [1.50 to 5.00] | 3.000 [0.50 to 4.50] | 4.250 [0.50 to 4.50] | 2.500 [0.50 to 8.00]
  D-PZQ | 3.000 [1.50 to 4.50] | 2.000 [1.00 to 4.50] | 3.500 [1.50 to 4.50] | 4.000 [0.50 to 4.50] | 4.500 [0.50 to 4.50] | 3.500 [0.50 to 8.00]
  racemate PZQ | 3.000 [1.50 to 4.50] | 1.750 [1.00 to 4.50] | 3.500 [1.50 to 4.50] | 3.500 [0.50 to 4.50] | 4.500 [0.50 to 4.50] | 2.500 [0.50 to 8.00]

4. Secondary Outcome: Apparent Terminal Half-life (t1/2) of L-PZQ, D-PZQ, and Racemate PZQ
Description: Apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50 percent in the final stage of its elimination.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: The PK population included all subjects who completed the study and for whom primary PK parameters could be calculated for the first two treatment periods. Here, "n" signifies those subjects who were evaluable for specified isomers (L-PZQ and D-PZQ) or the racemate mixture of PZQ for each arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 14 | 15
hours
  L-PZQ (n= 30,30,14,15,14,14) | 3.305 (49.1) | 3.830 (46.8) | 1.916 (72.2) | 4.202 (37.8) | 4.168 (34.9) | 3.072 (43.5)
  D-PZQ (n= 30,30,15,15,14,15) | 4.577 (34.7) | 4.618 (33.8) | 3.962 (37.2) | 4.346 (19.4) | 5.281 (30.1) | 4.347 (31.2)
  racemate PZQ (n= 30,30,15,15,14,15) | 4.462 (34.3) | 4.408 (35.8) | 3.775 (38.8) | 4.316 (24.4) | 4.889 (29.1) | 4.204 (30.2)

5. Secondary Outcome: Time Prior to the First Measurable (Non-zero) Concentration (Tlag) of L-PZQ, D-PZQ, and Racemate PZQ
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 14 | 15
hours
  L-PZQ | 0.000 [0.00 to 0.50] | 0.000 [0.00 to 0.50] | 0.000 [0.00 to 0.50] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  D-PZQ | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.50] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  racemate PZQ | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.50] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]

6. Secondary Outcome: AUC From Time Zero to the Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) Adjusted for the Actual Administered Dose (AUC0-t, Adj) of L-PZQ, D-PZQ, and Racemate PZQ
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 14 | 15
h*ng/mL
  L-PZQ | 1928.0 (47.4) | 1994.0 (61.1) | 300.5 (75.5) | 4770.1 (41.9) | 863.7 (70.2) | 1342.6 (86.0)
  D-PZQ | 7405.9 (28.2) | 8131.4 (39.0) | 2169.2 (46.7) | 14367.2 (34.0) | 4740.6 (56.5) | 6365.5 (41.5)
  racemate PZQ | 9476.3 (26.9) | 10266.0 (40.2) | 2515.2 (47.0) | 19262.2 (34.1) | 5694.0 (55.6) | 7929.9 (41.9)

7. Secondary Outcome: Extrapolated Area Under the Plasma Concentration Curve From Time Tlast to Infinity (AUCextra) of L-PZQ, D-PZQ, and Racemate PZQ
Description: AUCextra was reported in terms of percentage of AUC0-inf.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-inf
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 14 | 15
percentage of AUC0-inf
  L-PZQ (n= 30,30,14,15,14,14) | 1.86 (51.4) | 2.23 (66.3) | 5.25 (97.6) | 1.60 (79.9) | 5.52 (72.9) | 2.30 (63.7)
  D-PZQ (n= 30,30,15,15,14,15) | 1.30 (97.4) | 1.48 (90.4) | 2.26 (56.0) | 1.51 (106.9) | 3.69 (110.6) | 1.60 (97.6)
  racemate PZQ (n= 30,30,15,15,14,15) | 1.10 (101.0) | 1.24 (104.5) | 1.85 (59.0) | 1.38 (133.4) | 3.05 (117.2) | 1.38 (104.1)

8. Secondary Outcome: Apparent Terminal Elimination Rate Constant (λz) of L-PZQ, D-PZQ, and Racemate PZQ
Description: λz was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 14 | 15
1/h
  L-PZQ (n= 30,30,14,15,14,14) | 0.210 (49.1) | 0.181 (46.8) | 0.362 (72.2) | 0.165 (37.8) | 0.166 (34.9) | 0.226 (43.5)
  D-PZQ (n= 30,30,15,15,14,15) | 0.151 (34.7) | 0.150 (33.8) | 0.175 (37.2) | 0.159 (19.4) | 0.131 (30.1) | 0.159 (31.2)
  racemate PZQ (n= 30,30,15,15,14,15) | 0.155 (34.3) | 0.157 (35.8) | 0.184 (38.8) | 0.161 (24.4) | 0.142 (29.1) | 0.165 (30.2)

9. Secondary Outcome: Relative Bioavailability (Frel) of L-PZQ, D-PZQ, and Racemate PZQ
Description: Frel was calculated for Treatment A versus Treatment B only. It was calculated by using AUC0-∞, with treatment A as the Test and treatment B as the Reference. Frel = AUC0-inf (test) / AUC0-inf (reference).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent bioavailability
Groups:
- PZQ 40 mg/kg (Treatment A and Treatment B): Subjects who received a single oral dose of 40 mg/kg of test ODT-PZQ dispersed in water after a meal and reference PZQ formulation (Cysticide tablet) at a single dose of 40 mg/kg given with water orally after a meal in either of the four intervention periods.
Arm/Group | PZQ 40 mg/kg (Treatment A and Treatment B)
Number analyzed (Participants) | 30
percent bioavailability
  L-PZQ | 96.175 (46.70)
  D-PZQ | 90.951 (27.52)
  racemate PZQ | 92.2 (21.6)

10. Secondary Outcome: Apparent Total Body Clearance of Drug From Plasma (CL/f) of L-PZQ, D-PZQ, and Racemate PZQ
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 14 | 15
Liter/hour
  L-PZQ (n= 30,30,14,15,14,14) | 716.8 (45.0) | 691.3 (57.9) | 2028.4 (60.0) | 438.5 (45.8) | 1466.9 (60.6) | 971.1 (69.5)
  D-PZQ (n= 30,30,15,15,14,15) | 187.2 (33.3) | 170.7 (42.6) | 316.7 (47.6) | 145.5 (41.6) | 271.6 (62.8) | 227.6 (43.7)
  racemate PZQ (n= 30,30,15,15,14,15) | 293.3 (30.7) | 271.0 (42.6) | 548.7 (46.4) | 217.1 (41.0) | 455.6 (60.1) | 366.1 (43.2)

11. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/f) of L-PZQ, D-PZQ, and Racemate PZQ
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/f after oral dose was influenced by the fraction absorbed.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 14 | 15
Liters
  L-PZQ (n= 30,30,14,15,14,14) | 3417.6 (37.0) | 3820.4 (57.5) | 5605.6 (63.9) | 2658.4 (59.9) | 8820.4 (55.3) | 4304.4 (50.6)
  D-PZQ (n= 30,30,15,15,14,15) | 1236.0 (43.7) | 1137.4 (52.9) | 1810.1 (64.8) | 912.1 (40.0) | 2069.2 (70.5) | 1427.2 (41.5)
  racemate PZQ (n= 30,30,15,15,14,15) | 1887.7 (37.3) | 1723.7 (53.3) | 2987.7 (60.4) | 1352.0 (42.7) | 3213.2 (61.7) | 2220.2 (38.4)

12. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to Infinity (AUC0-inf) Adjusted for the Actual Administered Dose (AUC0-inf, Adj) of D-PZQ and Racemate PZQ
Description: AUC0-inf is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time. AUC0-inf, adj was defined as the AUC0-inf adjusted for the actual administered dose of D-PZQ and Racemate PZQ.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16 and 24 hours post-dose on Day 1 of each treatment
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 14 | 15
h*ng/mL
  D-PZQ | 7542.3 (29.2) | 8292.7 (39.4) | 2226.0 (46.1) | 14685.8 (35.5) | 4996.0 (58.5) | 6508.9 (41.8)
  racemate PZQ | 9627.2 (28.0) | 10446.9 (40.7) | 2569.5 (46.5) | 19679.5 (35.4) | 5956.0 (57.7) | 8091.8 (42.3)

13. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the stud drug.
Time Frame: Baseline up to end of treatment (up to Day 32)
Population: as for baseline characteristics
Measure: Number; unit: subjects
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 31 | 32 | 15 | 15 | 14 | 15
subjects
  TEAEs | 5 | 4 | 1 | 6 | 0 | 3
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0
  TEAE leading to Discontinuation | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Palatability Assessment Based on Visual Analog Scale (VAS) Score
Description: Palatability was assessed in terms of Flavor, Smell, Sweetness, Overall liking of the medicine, Taste and Acceptability to swallow, each parameter assessed on a 0 to 100 millimeter (mm) visual analog scale (VAS), where 0 indicates "Did not like" and 100 indicates "very much liked". Flavor, Smell, Sweetness and Overall liking of the medicine were evaluated immediately after taking the medication (Day 1, 0 Hour) and Taste and Acceptability to swallow were assessed 2-5 minutes post administration of medication.
Time Frame: Immediately and 2-5 minutes (min) after dosing on Day 1 of each treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millimiter (mm)
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 31 | 32 | 15 | 15 | 14 | 15
millimiter (mm)
  Day 1, 0 Hour: Flavour | 43.4 (30.25) | 44.6 (32.18) | 50.3 (32.24) | 46.1 (33.14) | 55.9 (31.20) | 20.1 (20.82)
  Day 1, 0 Hour: Smell | 60.7 (25.91) | 61.5 (24.57) | 47.5 (33.64) | 51.1 (26.11) | 51.7 (29.65) | 29.4 (29.34)
  Day 1, 0 Hour: Sweetness | 47.3 (27.12) | 41.2 (32.55) | 51.4 (31.91) | 50.7 (33.02) | 61.6 (21.19) | 12.9 (21.31)
  Day 1, 0 Hour: Overall liking | 46.8 (32.29) | 51.3 (30.67) | 50.2 (33.93) | 40.7 (31.60) | 48.8 (30.24) | 13.7 (20.07)
  Day 1, 2-5 Min After Medicine: Taste in Mouth | 39.7 (31.34) | 44.9 (30.74) | 44.7 (31.23) | 35.0 (32.21) | 46.7 (31.29) | 14.4 (21.07)
  Day1,2-5 Min After Medicine:Acceptable to Swallow | 68.2 (30.90) | 62.5 (26.48) | 55.7 (33.16) | 39.9 (33.71) | 61.1 (31.51) | 23.1 (29.19)

15. Secondary Outcome: Number of Subjects With Clinically Significant Change From Baseline in Vital Signs, Physical Examinations, Electrocardiogram (ECG) and Laboratory Parameters
Description: Vital signs included oral body temperature, blood pressure and pulse rate. Body weight was recorded for physical examinations. The 12-lead ECGs were recorded after the subjects have rested for at least 5 minutes in supine position. The parameters heart rate (HR), RR, PR, QRS, QT and QTcB calculated by the Bazett formula. Laboratory investigation including chemistry, hematology and urinalysis.
Time Frame: Baseline up to end of treatment (up to Day 32)
Population: as for baseline characteristics
Measure: Number; unit: subjects
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Number analyzed (Participants) | 31 | 32 | 15 | 15 | 14 | 15
subjects | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to end of treatment (up to Day 32)
Arm/Group | Treatment A: 40 mg/kg Test ODT-PZQ After Meal | Treatment B: 40 mg/kg Cysticide Tablet After Meal | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32 | 0/15 | 0/15 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 5/31 | 4/32 | 1/15 | 6/15 | 0/14 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: 40 mg/kg Test ODT-PZQ After Meal (N=31) | Treatment B: 40 mg/kg Cysticide Tablet After Meal (N=32) | Treatment C1: 20 mg/kg Test ODT-PZQ After Meal (N=15) | Treatment C2: 60 mg/kg Test ODT-PZQ After Meal (N=15) | Treatment D1: 40 mg/kg Test ODT-PZQ Without Meal (N=14) | Treatment D2: 40 mg/kg Cysticide Crushed Tablets After Meal (N=15)
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 4 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No